CLINICAL TRIAL: NCT05766241
Title: Investigating the Feasibility and Efficacy of a Novel Sensory-based Psychoeducation Program for Military Veterans With Posttraumatic Stress Disorder
Brief Title: Investigating a Novel Sensory-based Program for Veterans With PTSD
Acronym: SENSE-PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Veterans Affairs Canada (Unknown)
Responsible Party: Principal Investigator, Margaret McKinnon, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13743
Record Dates: First submitted 2022-09-28; First posted 2023-03-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: sensory; psychoeducation; Canadian Armed Forces; PTSD; virtual; veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a program group or a waitlist control group. Individuals in the waitlist control group will be offered the opportunity to participate in the program once they have completed the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program group (Experimental): Participants in this group will receive five weekly sessions of Sensory Strategies Training (SST), facilitated by a trained clinician or graduate/post-graduate student in a health-related field.
  Interventions: Behavioral: Sensory Strategies Training
- Waitlist control group (No Intervention): Participants in the waitlist control group will not receive SST or any other PTSD or sensory-processing treatments for the duration of the study.

INTERVENTIONS:
Behavioral: Sensory Strategies Training — In SST, participants will be introduced to the concept of sensory processing in the context of PTSD and will learn about the ways in which difficulties in this area can impact their affective, cognitive, and functional outcomes. Participants will learn about the effects of PTSD symptoms on their ability to regulate stressful situations and engage in social interactions, as well as the benefits of physical activity and proper sleep hygiene. Participants will also identify functional goals (e.g., reduce sensation-avoiding, better regulate physical and emotional reactions to trauma reminders, increase sensory sensitivity, etc.) which they will aim to achieve with the knowledge and resources gained from SST. Throughout the program, participants will learn various strategies to help with movement, sleep, and interacting with others, and will have opportunities to practice the strategies identified as being relevant to their specific needs during their baseline sensory assessment.
  Other Names: SST
  Arms: Program group

SUMMARY:
SENSE-PTSD is an randomized controlled trial (RCT) which will evaluate the feasibility and efficacy of a novel, sensory-based psychoeducational program for improving psychological, functional, sensory, and cognitive outcomes in Canadian military veterans with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a disorder that can happen after a person experiences an event that makes them feel extremely frightened or helpless (i.e., a traumatic event. Some examples of traumatic events include physical, sexual, or emotional abuse; automobile accidents; and military combat. Symptoms of PTSD typically include feeling overwhelmed by memories of the traumatic event, trying to avoid reminders of the traumatic event, feeling overly alert to danger, and experiencing difficulty regulating emotions. They can also include fluctuations in arousal in the body where one may feel high levels of arousal (e.g., increased heart rate, anxiety/stress, faster breathing) or low levels of arousal (e.g., decreased heart rate, numb, withdrawn). PTSD can hinder someone's ability to meet the demands of everyday life, including interacting with family, friends, and coworkers, which can in turn have negative consequences on their employment status, financial wellbeing, and bonds with others.

Engaging in military service can increase someone's risk for experiencing traumatic events. Examples of traumatic events commonly experienced by military personnel include severe injury, loss of life, and sexual misconduct (e.g., sexual harassment, gender discrimination), among others. While some treatments already exist for military personnel and veterans with PTSD, they tend to focus on the cognitive - or thought-based - symptoms of PTSD (e.g., gaps in memory, persistent negative thinking, difficulty with concentration and making plans), and can neglect physical or sensory regulation-based symptoms (e.g., muscle tension, shaking, crying, feeling restless, trouble sleeping).

This pilot study will examine a novel, virtual psychoeducational program called Sensory Strategies Training (SST). The main goal of this program is to provide military veterans with information and tools that they can use in their daily lives to reduce some of the PTSD symptoms mentioned above and expand the range of sensations they are able to tolerate, in effect increasing their overall ability to function in daily life. SST includes 5 one-on-one sessions with a trained clinician or graduate/post-graduate student in a mental health-related field, in which participants will learn about how PTSD symptoms may be affecting their lives and how to use sensory-based strategies to help reduce some of these symptoms. The main purpose of the current study is to inform our decision-making for a larger study that the investigators intend to conduct in the future. This larger study will explore how helpful SST is for improving PTSD symptoms in military veterans. The current pilot study will also explore this topic, but on a smaller scale.

Participants of the current study will be veterans of the Canadian Armed Forces (CAF; both active service and reservist) with PTSD. They will be randomized to either a psychoeducation program group, in which they will receive SST for 5 weeks, or a waitlist control group, in which they will receive no PTSD treatment for the same amount of time. Participants in the waitlist control group will be offered SST once they are finished participating in this study. The investigators will compare changes in self-reported PTSD symptoms and sensory processing before and after participants take part in SST or spend the equivalent amount of time on a waitlist to determine whether the program is effective. The investigators will also compare results 3 months later, to determine if the effects of the program are sustained over time. The study will be conducted entirely virtually via Zoom, an online video conferencing platform.

Ultimately, SST may be helpful for regulating the physiological and emotional functioning of military veterans with PTSD to help them tolerate a range of sensations, feelings, thoughts, and memories in the present moment. It is expected that the knowledge and skills gained from the sensory-based strategies will help participants identify and communicate their needs effectively and organize their behaviours in order to improve daily functioning, family relationships, and their engagement with the community.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults between the ages of 18 and 65
* Veterans of the Canadian Armed Forces (active service and/or reservist);
* Meet diagnostic criteria for PTSD on the Clinician Administered PTSD Scale (CAPS-5);
* Able to provide written informed consent;
* Have access to a smart phone, tablet, or computer with a working microphone and camera;
* Have access to consistent and reliable Internet.

Exclusion Criteria:

* Use benzodiazepines daily or almost daily;
* Use narcotics daily or almost daily;
* Diagnosis of substance use disorder in the past 3 months;
* History of severe head trauma with loss of consciousness or history of traumatic brain injury;
* History of neurological disorder;
* Diagnosis of a psychotic disorder or bipolar disorder;
* Diagnosis of a neurodevelopmental disorder;
* Have not had stable psychiatric medication for 6 months prior to study participation;
* Currently receiving counselling which targets trauma or sensory processing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate feasibility | 17 weeks
  Rate of recruitment per month.
Eligibility criteria feasibility | 17 weeks
  Percentage of individuals who are deemed eligible to participate in the study out of the total number of individuals who complete the pre-screening survey.
Length of completion of procedures feasibility | 17 weeks
  Time it takes to complete each study procedure.
Location logistics | 17 weeks
  Issues that arise as a result of the virtual nature of the study.
Attrition rates | 17 weeks
  Percentage of participants who drop out of SST.
Attendance rates of program | 17 weeks
  Percentage of SST sessions attended per participant.
Staff size feasibility | 17 weeks
  Facilitator feedback about how onerous their workload is.
Communication feasibility | 17 weeks
  Research team feedback on whether communication between research team members is adequate.

SECONDARY OUTCOMES:
Sensory difficulties | 17 weeks
  Changes in performance on the Adult/Adolescent Sensory Profile (semi-structured interview) at baseline, post-program, and 3-month follow-up. Scores can range between 60 and 300 with higher scores denoting greater sensory difficulties.
Occupational performance | 17 weeks
  Changes in performance on the Canadian Occupational Performance Measure (semi-structured interview) at baseline, post-program, and 3-month follow-up. Average performance and satisfaction scores are rated from 1 (poor performance/low satisfaction) to 10 (very good performance/high satisfaction). These scores are individually compared to prior scores at each time point (baseline, post-program and 3-month follow-up), with lower scores denoting greater sensory difficulties.
PTSD symptomatology (structured interview) | 17 weeks
  Changes in performance on Clinician Administered PTSD Scale (structured interview) at baseline, post-program, and 3-month follow-up. Scores can range between 0 and 120 with higher scores denoting more severe PTSD symptomatology.
Mental health symptomatology | 17 weeks
  Changes in performance on the Mini International Neuropsychiatric Interview (structured interview) at baseline, post-program, and 3-month follow-up. The Mini International Neuropsychiatric Interview will be used to indicate whether participants have PTSD or meet criteria for other psychiatric diagnoses. Diagnoses are made on a pass-or-fail basis, not reliant on minimum or maximum scores.
Depression, anxiety, and stress symptomatology | 17 weeks
  Changes in performance on Depression Anxiety Stress Scale 21-item version at baseline, post-program, and 3-month follow-up. Scores can range between 0 and 42 with higher scores denoting higher depression, anxiety, and/or stress symptomatology.
Dissociation | 17 weeks
  Changes in performance on the Multiscale Dissociation Inventory at baseline, post-program, and 3-month follow-up. Scores can range between 0 and 120 with higher scores denoting higher dissociative symptomatology.
PTSD symptomatology (checklist) | 17 weeks
  Changes in performance on the PTSD Checklist for DSM-5 at baseline, post-program, and 3-month follow-up. up. Scores can range between 0 and 80 with higher scores denoting higher PTSD symptomatology.
Emotion regulation | 17 weeks
  Changes in performance on the Difficulties in Emotion Regulation Scale at baseline, post-program, and 3-month follow-up. up. Scores can range between 36 and 180 with higher scores denoting poorer emotion regulation.
Sleep quality | 17 weeks
  Changes in performance on the Pittsburgh Sleep Quality Index at baseline, post-program, and 3-month follow-up. up. Scores can range between 0 and 21 with higher scores denoting poorer sleep quality.
Moral injury | 17 weeks
  Changes in performance on the Moral Injury Events Scale at baseline, post-program, and 3-month follow-up. up. Scores can range between 9 and 54 with lower scores denoting higher moral injury.
Verbal short-term/working memory | 17 weeks
  Changes in performance on the Digit Span neuropsychological assessments from the Wechsler Adult Intelligence Scales at baseline, post-program, and 3-month follow-up will be used to assess working memory. This task assesses working memory based on the average of digit sequences correctly remembered. Task difficulty dynamically varies based on the number of digits remembered, increasing or decreasing by 1 depending on whether the participants got the last trial correct. The test ends after 3 errors, with a maximum difficulty level of 25 and a minimum level of 2. The outcome measure is the maximum level achieved.
Attention | 17 weeks
  Changes in performance on the Feature Match neuropsychological assessment from the Wechsler Adult Intelligence Scales at baseline, post-program, and 3-month follow-up, will be used to assess attention. This task assesses attention based on one's ability to correctly identify similarities and differences between as many problems as possible within 90 seconds. The total score increases when participants respond correctly and decreases by the number of shapes in the current grid when participants respond incorrectly. The outcome measure is the total score.
Response inhibition | 17 weeks
  Changes in performance on the Double Trouble neuropsychological assessment from the Wechsler Adult Intelligence Scales at baseline, post-program, and 3-month follow-up, will be used to assess response inhibition. This task assesses response inhibition based on one's ability to make an appropriate response even when interference/distractors are present. To gain maximum points participants must solve as many problems as possible within 90 seconds, where the total score increases or decreases by 1 depending on if participants answer correctly or incorrectly. The outcome measure is the total score.
Executive functioning | 17 weeks
  Changes in performance on the Spatial Planning neuropsychological assessment from the Wechsler Adult Intelligence Scales at baseline, post-program, and 3-month follow-up, will be used to assess one's executive functioning. This task assesses executive functioning based on correctly solving specific problems in as few moves as possible within 3-minutes. After each trial, the total score is incremented by adding the minimum number of moves required multiplied by 2, minus the number of moves made. The outcome measure is the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McKinnon, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson CE, Ciarleglio MM, Aslan M, Marx BP, Ko J, Concato J, Proctor SP, Vasterling JJ. Associations Among Increases in Posttraumatic Stress Symptoms, Neurocognitive Performance, and Long-Term Functional Outcomes in U.S. Iraq War Veterans. J Trauma Stress. 2021 Jun;34(3):628-640. doi: 10.1002/jts.22663. Epub 2021 Mar 2. PMID 33650202
- [Background] Watkins LE, Sprang KR, Rothbaum BO. Treating PTSD: A Review of Evidence-Based Psychotherapy Interventions. Front Behav Neurosci. 2018 Nov 2;12:258. doi: 10.3389/fnbeh.2018.00258. eCollection 2018. PMID 30450043
- [Background] Regier DA, Kuhl EA, Kupfer DJ. The DSM-5: Classification and criteria changes. World Psychiatry. 2013 Jun;12(2):92-8. doi: 10.1002/wps.20050. PMID 23737408
- See also: McKinnon Trauma and Recovery Lab website — https://www.thetraumaandrecoverylab.com/